CLINICAL TRIAL: NCT01586104
Title: Cardiac-Sparing Whole Lung IMRT in Children and Young Adults With Lung Metastases: A Feasibility Study
Brief Title: Intensity-Modulated Radiation Therapy in Treating Younger Patients With Lung Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Kalapurakal, Attending Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lung IMRT; R21CA159547 (NIH)
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Adult Rhabdomyosarcoma; Lung Metastases; Metastatic Ewing Sarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Stage IV Adult Soft Tissue Sarcoma; Stage IV Wilms Tumor; Stage V Wilms Tumor; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma, Ewing; Sarcoma; Wilms Tumor | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (IMRT) (Experimental): Patients undergo cardiac-sparing whole lung intensity-modulated radiation therapy (IMRT).
  Interventions: Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: intensity-modulated radiation therapy — Undergo cardiac-sparing whole lung IMRT
  Other Names: IMRT

SUMMARY:
This pilot clinical trial studies intensity-modulated radiation therapy (IMRT) in treating younger patients with lung metastases. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To demonstrate the feasibility of delivering cardiac-sparing IMRT in a multi-institutional setting with central quality control for children and young adults with metastatic tumors in the lungs.

II. To prospectively determine the dosimetric advantages of whole lung IMRT treatment over standard whole lung irradiation by comparing treatment plans and different organ dose-volume histograms such as lungs, heart, thyroid gland, liver etc. in all patients enrolled in this study.

III. To determine the short-term efficacy (lung-metastases free survival) and acute tolerance of whole lung IMRT at a minimum period of six months after IMRT.

OUTLINE:

Patients undergo cardiac-sparing whole lung IMRT.

After completion of study treatment, patients are followed up for 1-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have a Wilms tumor, Ewing Sarcoma, Rhabdomyosarcoma or any other metastatic pediatric malignancy; patients may have a single or multiple pulmonary metastases at the time of diagnosis or at the time of recurrence; a pulmonary metastasis may be defined as one pulmonary nodule >= 1 cm or more than one pulmonary nodules >= 0.5 cm; a biopsy of the nodules may be considered in case of doubt
* The Karnofsky performance status must be >= 50 for patients > 16 years of age and the Lansky performance status must be >= 50 for patients =< 16 years of age
* Patients must not have received prior radiation therapy to any part of the thorax
* Adequate cardiac function defined as:
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram

  * Female patients of childbearing age must have a negative pregnancy test
  * Female patients who are lactating must agree to stop breast-feeding
  * Sexually active patients of childbearing potential must agree to use effective contraception

Exclusion Criteria:

* Patients enrolled on Children's Oncology Group protocols cannot be treated with whole lung IMRT on this study
* Patients who have a prior history of radiation therapy to the thorax or adjacent regions cannot be entered on this protocol
* Patient with Hodgkin's Lymphoma are not eligible for this study
* Patients with mediastinal masses or other pulmonary masses requiring additional mediastinal or lung irradiation beyond the whole lung irradiation (WLI) doses stated in this protocol are ineligible for this study
* Patients who may require concurrent or sequential irradiation to sites beyond the chest such as the neck, flank, abdomen or liver are eligible for this study

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walterhouse, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (7):
- United States (7):
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Ann & Rober H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (IMRT): Patients undergo cardiac-sparing whole lung IMRT.
  intensity-modulated radiation therapy: Undergo cardiac-sparing whole lung IMRT
Period: Overall Study
Arm/Group | Treatment (IMRT)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (IMRT)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 13 [1 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Delivering Cardiac-sparing IMRT With Central Quality Control in 20 Subjects
Description: Feasibility is defined as an enrolled patient receiving the IMRT treatment as stipulated in the protocol. Feasibility of delivering whole lung IMRT will be demonstrated by obtaining central (Quality Assurance Review Center 'QARC') quality control approval of enrolled patient treatment plans according to the protocol guidelines for the 20 subjects enrolled onto the study. If an enrolled patient did not receive the IMRT treatment as stipulated in the protocol this subject then the treatment will be considered not feasible in this patient.
Time Frame: All IMRT treatment plans were centrally reviewed within 1-2 days of receipt of the radiation therapy plan. The feasibility was determined as 'feasible' if deemed in accordance with protocol guidelines after central QARC review within 1-2 days of receipt.
Population: 14 patients had pediatric sarcomas; 5 had Wilms tumor; 1 had hepatoblastoma. 15/20 received RT to primary site. 15 had CS-IMRT as part of primary therapy vs 5 had CS-IMRT at relapse/progressive disease. At time of CS-IMRT, 18/20 patients' lung tumors were in remission/stable & 2 had progressive disease.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (IMRT): Patients had radiation therapy planning performed for cardiac-sparing whole lung intensity-modulated radiation therapy (IMRT) according to stipulated guidelines in the protocol.
Arm/Group | Treatment (IMRT)
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: Short-term Efficacy (Lung-metastases Free Survival, Overall Survival, Pulmonary Relapse, Deceased From Progressive Disease)
Description: Serial CT scans of the chest were examined to determine lung-metastasis free survival
Time Frame: From date of enrollment until the date of first documented progression, relapse or date of death from any cause up to an average of 3 years.
Population: Overall survival and incidence rates of additional relevant clinical data
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (IMRT)
Number analyzed (Participants) | 20
Participants
  2yr overall survival | 18
  3yr overall survival | 18
  2yr lung-metastasis progression free survival | 13
  3yr lung-metastasis progression free survival | 10
  Pulmonary relapse | 8
  Pulmonary relapse - after primary therapy: number analyzed (Participants) | 15
  Pulmonary relapse - after primary therapy | 4
  Pulmonary relapse - after relapse/progression: number analyzed (Participants) | 5
  Pulmonary relapse - after relapse/progression | 4
  Deceased from progressive disease | 2

3. Secondary Outcome: Mean Percentage Radiation Dose to Organ Volumes
Description: The IMRT and standard anteroposterior (AP-PA) treatment plans were reviewed and compared for target coverage and organ dose-volume histograms. The mean percentage volume of the organ or organ sub-region receiving a percentage of the dose was estimated from the computerized treatment plans for these two techniques were estimated and compared statistically
Time Frame: This outcome is measured from central review of radiation plans within 1-2 days of receipt.
Measure: Mean (Standard Deviation); unit: Mean % radiation dose to % organ volume
Arm/Group | Treatment (IMRT)
Number analyzed (Participants) | 20
Mean % radiation dose to % organ volume
  Heart - V50 (%) for IMRT | 96 (5.4)
  Heart - V50 (%) for AP- PA | 100 (0.8)
  Heart - V83 (%) for IMRT | 65 (12.1)
  Heart - V83 (%) for AP-PA | 100 (2.2)
  Heart - V95 (%) for IMRT | 39 (15.5)
  Heart- V95 (%) for AP-PA | 97 (6.7)
  Left Ventricle - V50 (%) for IMRT | 95 (7.8)
  Left Ventricle - V50 (%) for AP-PA | 100 (0)
  Left Ventricle - V95 (%) for IMRT | 33 (15.9)
  Left Ventricle - V95 (%) for AP-PA | 99 (2.7)
  Right Ventricle - V50 (%) for IMRT | 91 (9.8)
  Right Ventricle - V50 (%) for AP-PA | 100 (1.6)
  Right Ventricle - V83 (%) for IMRT | 42 (12.7)
  Right Ventricle - V83 (%) for AP-PA | 99 (4)
  Right Ventricle - V95 (%) for IMRT | 18 (8.9)
  Right Ventricle - V95 (%) for AP-PA | 97 (8.2)
  Right Atrium - V50 (%) for IMRT | 99 (0.4)
  Right Atrium - V50 (%) for AP-PA | 99 (0.7)
  Right Atrium - V95 (%) for IMRT | 57 (22.5)
  Right Atrium - V95 (%) for AP-PA | 97 (11.1)
  Left Atrium V50 (%) for IMRT | 99 (0.4)
  Left Atrium V50 (%) for AP-PA | 100 (0.2)
  Left Atrium - V95 (%) for IMRT | 55 (22.3)
  Left Atrium - V95 (%) for AP-PA | 94 (15.4)
  Right Coronary Artery - V95 (%) for IMRT | 100 (0)
  Right Coronary Artery - V95 (%) for AP-PA | 100 (0)
  Left Coronary Artery - V95 (%) for IMRT | 88 (9.9)
  Left Coronary Artery - V95 (%) for AP-PA | 99 (1.3)
  Myocardium - V50 (%) for IMRT | 94 (8)
  Myocardium - V50 (%) for AP-PA | 100 (0)
  Myocardium - V95 (%) for IMRT | 69 (7.56)
  Myocardium - V95 (%) for AP-PA | 99 (0.88)
  Thyroid - V50 (%) for IMRT | 44 (32.5)
  Thyroid - V50 (%) for AP-PA | 33 (31.3)
  Kidneys - V50 (%) for IMRT | 5 (7.6)
  Kidneys - V50 (%) for AP-PA | 6 (6.8)
  Stomach - V50 (%) for IMRT | 62 (21.7)
  Stomach - V50 (%) for AP-PA | 62 (24.5)
  Liver - V50 (%) for IMRT | 55 (11.4)
  Liver - V50 (%) for AP-PA | 54 (11.4)
Statistical Analysis 1: Comparison: Treatment (IMRT); Feasibility will be defined as an enrolled patient receiving the IMRT treatment as planned. It is expected that the treatment will be feasible in at least 90% of patients. If the treatment is feasible in 16 or more out of 20 patients, then the treatment will be declared feasible. If the true feasibility rate is 90%, then there is a 4.3% chance that 15 or fewer feasible patients will be observed; Test type: Other — With 20 patients, there is 80% power to detect a difference of 100% with Standard lung RT versus 93% with IMRT assuming a standard deviation of 8 (as seen for the whole heart), a one tailed test and a Bonferroni correction for 4 statistical tests so that each test is done at p<0.0125; p < 0.0125, Bonferroni corrected at p<0.0125 — The reported p value was calculated. The statistical analysis performed is attached to the outcome measure reported; Lung-metastases-free survival will be estimated using Kaplan-Meier survival curves (minimum period of six months)

ADVERSE EVENTS:
Arm/Group | Treatment (IMRT)
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (IMRT) (N=20)
Deceased from progressive disease. (General disorders) | 2 (2) — Multi-organ failure from progressive and terminal cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes